CLINICAL TRIAL: NCT05851560
Title: Post-thyroid Surgery Adhesion Prevention Using Oxidized Regenerated Cellulose and Hyaluronic Acid: Prospective, Single-blinded, Randomized Study
Brief Title: Prospective Comparison of the Effect on Antiadhesive Barriers During Thyroid Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 202111057DINB; NTUH 113-CTC0004 (Other Grant/Funding Number: National Taiwan University Hospital)
Record Dates: First submitted 2023-04-17; First posted 2023-05-09 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Thyroidectomy; Goiter; Thyroid Cancer
MeSH Terms: conditions — Goiter; Thyroid Neoplasms | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): control group that does not use antiadhesive material
- Oxidized regenerated cellulose(ORC) Group (Experimental): The group that uses Oxidized regenerated cellulose(ORC) as antiadhesive material during thyroid surgery.
  Interventions: Drug: Oxidized regenerated cellulose(ORC)
- Hyaluronic acid(HA) Group (Experimental): The group that uses Hyaluronic acid(HA) as antiadhesive material during thyroid surgery.
  Interventions: Drug: Hyaluronic acid(HA)

INTERVENTIONS:
Drug: Oxidized regenerated cellulose(ORC) — Investigate the antiadhesive effect of multiple antiadhesive barriers in thyroid surgery
  Other Names: Anti-Adhesion Agent
  Arms: Oxidized regenerated cellulose(ORC) Group
Drug: Hyaluronic acid(HA) — Hyaluronic acid(HA)
  Other Names: Anti-Adhesion Agent
  Arms: Hyaluronic acid(HA) Group

SUMMARY:
Despite use of meticulous surgical techniques and regardless of surgical access via conventional open or endoscopy, postoperative adhesions develop in the vast majority of patients undergoing neck surgery. Such adhesions represent not only adhesion reformation at sites of adhesiolysis, but also de novo adhesion formation at sites of surgical procedures. Improved understanding of the pathophysiology of adhesion development and distinguishing variations in the molecular biologic mechanisms represent future opportunities to improve the reduction of postoperative adhesions.

After surgical tissue injury, there were local release of histamine, cytokines, and growth factors that lead to adhesion development. Other than survival or safety issues, cosmetics concerns and quality of life are the motifs after thyroid surgeries currently. Pos-thyroidectomy adhesions include various symptoms such as neck discomfort, neck tightness, skin adhesion to the trachea, skin scarring from adhesive reaction, and vocal cord palsy or impairment of laryngeal vertical movement. Relief of the adhesion through wound massage or anti-adhesion agents could reduce neck discomfort and voice changes.Although oxidized regenerated cellulose (ORC) and hyaluronic acid (HA) appeared to be safe and effective to decrease the incidence of adhesions, to improve adhesion-related neck discomfort, and to prevent skin adhesion to the trachea after neck surgery. The application of antiadhesive barriers after neck surgery is safe but the effect is still uncertain. Thus, we aim to confirm the antiadhesive effect of multiple antiadhesive barriers in thyroid/parathyroid surgery.

DETAILED DESCRIPTION:
The postsurgical adhesions remain a significant cause of morbidity for a large number of patients in thyroid and parathyroid surgeries, despite use of meticulous surgical techniques and regardless of surgical access via conventional open or endoscopy. Such adhesions represent not only adhesion reformation at sites of adhesiolysis, but also de novo adhesion formation at sites of surgical procedures. A number of products, in the form of film or fluid, are used to prevent postoperative adhesion formation. These products normally serve as barriers to separate the contact of the damaged tissue surfaces in many animal models and some clinical practices. However, there are few evidences for surgeons to use or no use, or choose the suitable products in their clinical practice in neck surgeries. Improved understanding of the pathophysiology of adhesion development and distinguishing variations in the molecular biologic mechanisms represent future opportunities to improve the reduction of postoperative adhesions.

After surgical tissue injury, there were local release of histamine, cytokines, and growth factors that lead to adhesion development . Local tissue inflammation processes initiate capillary leakage of serosanguineous fluid including clotting factors, and recruitment of macrophages and other cells, including fibroblasts. Cutting, fulguration, ligation of the macrovasculature and microvasculature leads to a state of tissue hypoxemia. Along with the accumulation of metabolic byproducts such as lactic acid, the lowering the pH of the injured tissue, and the conversion from aerobic to anaerobic metabolism within the injured tissues. Tissue hypoxia also results in creation of oxidative stress, with production of oxygen and nitrogen free radicals, which can result in DNA mutations, alterations of mitochondrial DNA, and generation of oxidized proteins.

Subsequently induce lipid peroxidation and protein nitration. The known factors involved in the inflammatory-like response that lead to adhesion development, are type 1 collagen, transforming growth factor b1 (TGF-b1), tumor necrosis factor a (TNF-a), interleukin 6 (IL-6), and vascular endothelial growth factor (VEGF). Of note, the scavenging of free radicals such as superoxide by superoxide dismutase can prevent the development of the adhesion phenotype . Other processes affected include plasminogen activator activity (PAA) (a function of tissue plasminogen activator and its inhibitor, plasminogen activator inhibitor-1), metalloproteinase activity, and extracellular matrix deposition (such as collagen 1, collagen 3, and fibronectin). There is also initiation of processes leading to angiogenesis, which can lead to new vessel formation that could resupply oxygen to these tissues as well as remove metabolic byproducts.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20 years of age.
* Patients diagnosed with benign goiter or thyroid cancer that will undergo open thyroidectomy (either unilateral or bilateral total thyroidectomy with or without central lymph node dissection).
* Naïve patients to thyroid surgery.
* Subjects are willing to comply with all aspects of the study and have signed informed consent form.

Exclusion Criteria:

* Pregnant or lactating female patients.
* Presence of severe and uncontrolled illness such as stroke, hypertension, diabetes, chronic renal failure, coagulopathy.
* Concurrent diseases/conditions which will be unable to evaluate the outcomes.
* Patients with previous neck radiotherapy within 1 year.
* Patients receiving any adhesion prevention adjuvant.
* Previous history of Keloid or hypertrophic scar.
* Participate are hypersensitive to anti-adhesion agents.
* Participate in another clinical trial within 1 month.
* Participate have drug or alcohol abuse.
* Patients' presence of surgical site infection or uncontrolled bleeding.
* Anticoagulant used within a week from surger

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Chinese version of Dysphagia Handicap Index(DHI) | pre-operation
  Evaluate the swallowing difficulty
Chinese version of Dysphagia Handicap Index(DHI) | post-operation(week 2)
  Evaluate the swallowing difficulty
Chinese version of Dysphagia Handicap Index(DHI) | post-operation( month1)
  Evaluate the swallowing difficulty
Chinese version of Dysphagia Handicap Index(DHI) | post-operation(month 6)
  Evaluate the swallowing difficulty
Chinese version of Dysphagia Handicap Index(DHI) | post-operation( month12)
  Evaluate the swallowing difficulty

SECONDARY OUTCOMES:
Adhesion severity | post-operation(week 2)
  Evaluate the adhesion severity by using questionnaires
Adhesion severity | post-operation(month1)
  Evaluate the adhesion severity by using questionnaires
Adhesion severity | post-operation(month 6)
  Evaluate the adhesion severity by using questionnaires
Adhesion severity | post-operation(month12)
  Evaluate the adhesion severity by using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hsun Wu, Study Chair — MD，PhD
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuo TC, Chen KY, Tsai YJ, Lin MT, Chang CH, Wu MH. Post-thyroid surgery adhesion prevention using oxidized regenerated cellulose and hyaluronic acid: prospective, single-blinded, randomized study. BJS Open. 2025 Jul 1;9(4):zraf079. doi: 10.1093/bjsopen/zraf079. PMID 40613790